CLINICAL TRIAL: NCT04494776
Title: Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-COV-2) Infection (COVID-19) in Kidney Transplant Recipients: a Brazilian Multicenter Study
Brief Title: SARS-COV-2 Infection in Kidney Transplant Recipients: a Brazilian Multicenter Study
Status: Recruiting | Type: Observational
Sponsor: Helio Tedesco Silva Junior (Other)
Collaborators: Hospital do Rim e Hipertensão (Other)
Responsible Party: Sponsor-Investigator, Helio Tedesco Silva Junior, Principal Investigator, Hospital do Rim e Hipertensão
Organization: Hospital do Rim e Hipertensão (Other)
Other Study IDs: 30631820.0.1001.8098
Record Dates: First submitted 2020-07-16; First posted 2020-07-31 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: SARS-CoV-2 Infection; Kidney Transplant Infection
Keywords: SARS-CoV-2 Infection; Kidney Transplant Infection; Kidney Transplant
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
COVID-19 is the pandemic disease caused by the SARS-CoV-2 coronavirus. It is a highly contagious viral disease, the condition of which main clinical symptoms are characterized by fever and respiratory symptoms. Evidence indicates to worse outcomes in patients with pre-existing diseases, such as diabetes, arterial hypertension, heart disease, pneumopathies, chronic kidney disease, and immunodeficiencies. Recipients of kidney transplants make prolonged use of immunosuppressive drugs to inhibit the acquired immune response, notably the activity of lymphocytes. Due to this potential to modulate the immune and inflammatory response, it is speculated that the clinical and laboratory condition of COVID-19 in these patients is atypical. Preliminary evidence suggests worse outcomes of COVID-19 in immunosuppressed patients, as carriers of cancer. However, information on kidney transplant recipients is insufficient. So far, only reports of the case are available in the literature with different clinical presentations and outcomes. The aim of this study is, therefore, to characterize the demographics, clinical and laboratory conditions, and the outcomes of COVID-19 in kidney transplant recipients in a national multicenter cohort.

DETAILED DESCRIPTION:
COVID-19 is the pandemic disease caused by the SARS-CoV-2 coronavirus. It is a highly contagious viral disease, the condition of which main clinical symptoms are characterized by fever and respiratory symptoms. Evidence indicates to worse outcomes in patients with pre-existing diseases, such as diabetes, arterial hypertension, heart disease, pneumopathies, chronic kidney disease, and immunodeficiencies. Recipients of kidney transplants make prolonged use of immunosuppressive drugs to inhibit the acquired immune response, notably the activity of lymphocytes. Due to this potential to modulate the immune and inflammatory response, it is speculated that the clinical and laboratory condition of COVID-19 in these patients is atypical. Preliminary evidence suggests worse outcomes of COVID-19 in immunosuppressed patients, as carriers of cancer. However, information on kidney transplant recipients is insufficient. So far, only reports of the case are available in the literature with different clinical presentations and outcomes. The aim of this study is, therefore, to characterize the demographics, clinical and laboratory conditions (mechanical ventilation, need for dialysis, need for ICU admission during evolution) and the outcomes of COVID-19 (death and graft loss within 3 months after infection up to 3 months after resolution) in kidney transplant recipients in a national multicenter cohort.Inclusion Criteria:1. Kidney transplant recipients, which may be multi-organ recipients, transplanted in any follow-up period; 2. Positive diagnostic test for COVID-19 (detection of viral load, test for detection of antigens or tests for detection of antibodies); 3.Outpatient or hospital management; 4.Adults and children. Exclusion Criteria: None

ELIGIBILITY:
Inclusion Criteria:

1. Kidney transplant recipients, which may be multi-organ recipients, transplanted in any follow-up period;
2. Positive diagnostic test for COVID-19 (detection of viral load, test for detection of antigens or tests for detection of antibodies);
3. Outpatient or hospital management;
4. Adults and children.

Exclusion Criteria:

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: COVID-19 kidney transplant recipients confirmed by diagnostic test.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2020-05-21 (Actual); Primary Completion 2022-12-03 (Actual); Study Completion 2025-04-02 (Estimated)

PRIMARY OUTCOMES:
Death | Up to 3 months after resolution
  Death within 3 months after infection (Yes/No).
Graft loss | Up to 3 months after resolution
  Graft loss up to 3 months after infection (Yes/No).

SECONDARY OUTCOMES:
Hospitalization | Until discharge date, an average of 1 month
  Composite outcomes: Mechanical ventilation (Yes/No); Need for dialysis (Yes/No); Need for ICU admission during evolution (Yes/No).

CONTACTS AND LOCATIONS:
Overall Officials: Jose Osmar Medina, Study Director — Hospital do Rim
Locations (1):
- Hospital do Rim, São Paulo, Aão Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Conti P, Ronconi G, Caraffa A, Gallenga CE, Ross R, Frydas I, Kritas SK. Induction of pro-inflammatory cytokines (IL-1 and IL-6) and lung inflammation by Coronavirus-19 (COVI-19 or SARS-CoV-2): anti-inflammatory strategies. J Biol Regul Homeost Agents. 2020 March-April,;34(2):327-331. doi: 10.23812/CONTI-E. PMID 32171193
- [Background] D'Antiga L. Coronaviruses and Immunosuppressed Patients: The Facts During the Third Epidemic. Liver Transpl. 2020 Jun;26(6):832-834. doi: 10.1002/lt.25756. Epub 2020 Apr 24. No abstract available. PMID 32196933
- [Background] Liang W, Guan W, Chen R, Wang W, Li J, Xu K, Li C, Ai Q, Lu W, Liang H, Li S, He J. Cancer patients in SARS-CoV-2 infection: a nationwide analysis in China. Lancet Oncol. 2020 Mar;21(3):335-337. doi: 10.1016/S1470-2045(20)30096-6. Epub 2020 Feb 14. No abstract available. PMID 32066541
- [Background] Zhu L, Xu X, Ma K, Yang J, Guan H, Chen S, Chen Z, Chen G. Successful recovery of COVID-19 pneumonia in a renal transplant recipient with long-term immunosuppression. Am J Transplant. 2020 Jul;20(7):1859-1863. doi: 10.1111/ajt.15869. Epub 2020 Mar 31. PMID 32181990
- [Background] Guillen E, Pineiro GJ, Revuelta I, Rodriguez D, Bodro M, Moreno A, Campistol JM, Diekmann F, Ventura-Aguiar P. Case report of COVID-19 in a kidney transplant recipient: Does immunosuppression alter the clinical presentation? Am J Transplant. 2020 Jul;20(7):1875-1878. doi: 10.1111/ajt.15874. Epub 2020 Apr 9. PMID 32198834
- [Derived] Modelli de Andrade LG, de Sandes-Freitas TV, Requiao-Moura LR, Viana LA, Cristelli MP, Garcia VD, Alcantara ALC, Esmeraldo RM, Abbud Filho M, Pacheco-Silva A, de Lima Carneiro ECR, Manfro RC, Costa KMAH, Simao DR, de Sousa MV, Santana VBBM, Noronha IL, Romao EA, Zanocco JA, Arimatea GGQ, De Boni Monteiro de Carvalho D, Tedesco-Silva H, Medina-Pestana J; COVID-19-KT Brazil. Development and validation of a simple web-based tool for early prediction of COVID-19-associated death in kidney transplant recipients. Am J Transplant. 2022 Feb;22(2):610-625. doi: 10.1111/ajt.16807. Epub 2021 Sep 2. PMID 34416075